CLINICAL TRIAL: NCT06439407
Title: An Open-label, Randomized, Controlled, Exploratory Clinical Trial to Preliminarily Assess the Safety and Feasibility of SAT-014, a Software for Alleviating Symptoms of Trauma and Stress-related Disorders
Brief Title: Clinical Trial to Preliminarily Assess the Safety and Feasibility of SAT-014, a Software for Alleviating Symptoms of Trauma and Stress-related Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S-Alpha Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAT014-KP-001
Record Dates: First submitted 2024-05-27; First posted 2024-06-03 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-08

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAT-014 (Experimental)
  Interventions: Device: SAT-014(Software as Medical Device)
- Maintain previous treatment (Other)
  Interventions: Device: SAT-014(Software as Medical Device)

INTERVENTIONS:
Device: SAT-014(Software as Medical Device) — SAT-014(Software as Medical Device) + maintain previous treatment

SUMMARY:
Failure to adapt to stress leads to functional impairments in various areas, including social, occupational, educational, and other significant domains, necessitating therapeutic intervention. Interventions through mobile app in the form of software can provide a new alternative for alleviating symptoms caused by psychological trauma by increasing accessibility to early intervention for trauma patients. This study aims to preliminarily assess the safety and feasibility of a psychological traum intervention by developing SAT-014 to help patients with trauma and stress-related disorder continue effective treatment in a stable environment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (19 years and older)
2. Have experienced clinically significant psychological trauma within the 6 months prior to screening visit
3. Met the diagnostic criteria for Post-Traumatic Stress Disorder (PTSD) or Adjustment Disorder (AD) category as evaluated by MINI (Mini-International Neuropsychiatric Interview)
4. Score between 17 and 38 points on the IES-R (Impact of Event Scale-Revised)
5. Score of 4 or less on CGI (Clinical Global Impression)
6. Capable of complying the activity instructions provided the app

Exclusion Criteria:

1. Have been diagnosed with schizophrenia, bipolar disorder, and psychotic disorder
2. Have been diagnosed with neurodevelopmental disorder, neurocognitive disorder, or organic mental disorder
3. Severe depression (PHQ-9 score of 20 or greater)
4. Comorbid with severe personality disorder
5. Diagnosed with substance use disorder excluding nicotine and caffeine and with severe alcohol use disorder
6. Have made a suicide attempt within 3 months and are judged to be at high risk for suicide by a psychiatrist
7. Pregnant or lactating
8. Currently participating in another clinical trial or have participated in another trial within 90 days from screening
9. Others deemed unsuitable for participation in this clinical trial at the discretion of the investigator due to ethical concerns or potential impact on the trial outcome

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Change in IES-R (Impact Event Scale-Revised) score | Baseline, 3weeks, 6weeks, 10weeks
  The Korean version of the Impact Event Scale-Revised (IES-R) consists of 22 items each rated on a 5-point scale ranging from 0 to 4. The total score ranges from 0 to 88, with higher scores indicating a greater risk of post-traumatic stress disorder and a worse outcome.
Change in PCL-5 (PTSD Checklist-5) score | Baseline, 3weeks, 6weeks, 10weeks
  The PTSD Checklist for DSM-5 (PCL-5) consists of 20 items, each rated on a scale from 0 to 4. The total score ranges from 0 to 80, with higher scores indicating greater distress due to symptoms related to past stressful experiences and a worse outcome.
Change in GAD-7 (Generalized Anxiety Disorder 7 item scale) score | Baseline, 3weeks, 6weeks, 10weeks
  The Generalized Anxiety Disorder 7-item scale (GAD-7) consists of 7 items, each rated on a scale from 0 to 3. The total score ranges from 0 to 21, with higher scores indicating more severe anxiety symptoms and a worse outcome.
Change in BAI (Beck Anxiety Inventory) score | Baseline, 3weeks, 6weeks, 10weeks
  The Beck Anxiety Inventory (BAI) consists of 21 items, each rated on a scale from 0 to 3. The total score ranges from 0 to 63, with higher scores indicating more severe anxiety symptoms and a worse outcome.
Change in PHQ-9 (Patient Health Questionnaire-9; depression screening tool) score | Baseline, 3weeks, 6weeks, 10weeks
  The Patient Health Questionnaire-9 (PHQ-9) consists of 9 items, each rated on a scale of 0 to 3. The total score ranges from 0 to 27, with higher scores indicating more severe symptoms and a worse outcome.
Change in QIDS-SR (Quick Inventory of Depressive Symptomatology-Self Report) score | Baseline, 3weeks, 6weeks, 10weeks
  The Quick Inventory of Depressive Symptomatology-Self Report (QIDS-SR) consist of 16 items, each rated on a scale of 0 to 3. It evaluates responses to 16 items based on criteria for nine depressive symptoms. The total score ranges from 0 to 27, with higher scores indicating more severe symptoms and a worse outcome.
Change in CGI (Clinical Global Impression) score | Baseline, 3weeks, 6weeks, 10weeks
  The CGI consists of two items: (a) the clinician's overall impression of the patient's severity of illness and (b) global improvement over time. The severity of illness is rated on a scale from 1 to 7, with a higher score indicating more severe illness and a worse outcome. Global improvement is also rated on a scale from 1 to 7, with a higher score indicating a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea